CLINICAL TRIAL: NCT07287995
Title: A Phase 1b/2 Study of ASP2998 as Monotherapy and in Combination With Standard Therapies in Participants With Locally Advanced Unresectable or Metastatic Solid Tumors
Brief Title: A Study of ASP2998 Given by Itself and Given With Standard Therapies in People With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2998-CL-0101; 2025-524567-21 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Malignant Solid Tumors
Keywords: ASP2998; Safety; Tolerability; Pembrolizumab; Enfortumab Vedotin; Carboplatin; Non-small cell lung cancer; Gastroesophageal junction cancer; Breast cancer; Pharmacokinetics; Urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Carcinoma, Transitional Cell | interventions — pembrolizumab; enfortumab vedotin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ASP2998 Dose Escalation (Experimental): Participants with urothelial carcinoma (UC), NSCLC, gastric/GEJ cancer or breast cancer (HER2-negative) will receive sequential doses of ASP2998 in a 21-day cycle.
  Interventions: Drug: ASP2998
- ASP2998 Dose Expansion (Experimental): Participants with UC or NSCLC will receive ASP2998 in a 21-day cycle with dose level(s) selected from dose escalation.
  Interventions: Drug: ASP2998
- ASP2998 Monotherapy Dose Escalation (Tumor Specific) (Experimental): Participants with select tumor types will receive ASP2998 in a 21-day cycle at dose level(s) based on emerging data.
  Interventions: Drug: ASP2998
- ASP2998 Monotherapy Dose Expansion (Tumor Specific) (Experimental): Participants with select tumor types will receive ASP2998 in a 21-day cycle at dose level(s) based on emerging data.
  Interventions: Drug: ASP2998
- ASP2998 Combination Therapy Dose Escalation (Tumor Specific) (Experimental): Participants with select tumor types will receive ASP2998 in a 21-day cycle at dose level(s) based on emerging data.
  Interventions: Drug: ASP2998; Drug: Pembrolizumab; Drug: Enfortumab Vedotin; Drug: Carboplatin
- ASP2998 Combination Therapy Dose Expansion (Tumor Specific) (Experimental): Participants with select tumor types will receive ASP2998 in a 21-day cycle at dose level(s) based on emerging data.
  Interventions: Drug: ASP2998; Drug: Pembrolizumab; Drug: Enfortumab Vedotin; Drug: Carboplatin

INTERVENTIONS:
Drug: ASP2998 — Intravenous infusion
Drug: Pembrolizumab — Intravenous infusion
  Other Names: Keytruda
  Arms: ASP2998 Combination Therapy Dose Escalation (Tumor Specific); ASP2998 Combination Therapy Dose Expansion (Tumor Specific)
Drug: Enfortumab Vedotin — Intravenous infusion
  Other Names: Padcev
  Arms: ASP2998 Combination Therapy Dose Escalation (Tumor Specific); ASP2998 Combination Therapy Dose Expansion (Tumor Specific)
Drug: Carboplatin — Intravenous infusion
  Arms: ASP2998 Combination Therapy Dose Escalation (Tumor Specific); ASP2998 Combination Therapy Dose Expansion (Tumor Specific)

SUMMARY:
Specific proteins found in tumors help the tumors spread and grow. People with solid tumors often have a protein called TROP2 in their tumor. ASP2998 is being developed to attach to TROP2 and then attack the tumor cells in people with solid tumors. ASP2998 will either be given by itself, or given together with one or more of standard cancer treatments pembrolizumab, carboplatin, and enfortumab vedotin.

This is an early development study to collect information about ASP2998 in people with solid tumors. In this study ASP2998 will be given to humans for the first time. Early development studies are mostly about safety, but also to find the most suitable dose. Other aims are to check if ASP2998 shows signs of reducing tumor growth, to learn how the body processes ASP2998, and to check if there are changes either in the TROP2 protein or in the immune system.

The main aim of the study is to check the safety of ASP2998 when given by itself and given with the standard cancer treatments, and how well it is tolerated.

People in this study will be adults with locally advanced, unresectable or metastatic solid tumors. Locally advanced means the cancer has spread to nearby tissue. Unresectable means the cancer cannot be removed by surgery. Metastatic means the cancer has spread to other parts of the body. People's cancer came back or became worse after previous treatment or they couldn't receive treatment. Some people who had previously refused treatment may be able to take part. This will depend on which study treatment they receive.

People will either have cancer in the bladder lining (urothelial cancer), non-small cell lung cancer (NSCLC), gastric cancer or cancer where the food pipe joins the stomach (gastroesophageal cancer, or GEJ), or certain types of breast cancer.

People cannot take part if the cancer cells have spread to the thin tissue covering the brain and spinal cord (leptomeningeal disease), have symptoms of cancer in the brain or nervous system, or need medicines to suppress their immune system.

In this study, ASP2998 will be given to humans for the first time. ASP2998 will either be given by itself, or given together with one or more of standard cancer treatments pembrolizumab, carboplatin and enfortumab vedotin. The standard cancer treatment given will depend on which cancer people have.

The study will have 2 parts.

In Part 1, different small groups of people will receive lower to higher doses of ASP2998 given by itself or together with one or more of the standard cancer treatments. Any medical problems will be recorded for each dose. This is done to find suitable doses of ASP2998 to use in Part 2.

In Part 2, other different small groups will receive suitable doses of ASP2998 worked out from Part 1. ASP2998 will either be given by itself or given together with one or more of the standard cancer treatments. This part will also check how each type of cancer responds to ASP2998 when given by itself or together with the standard cancer treatments.

In both parts of the study, safety checks will be done at each visit, and the doctors will continue to check for medical problems throughout the study. ASP2998 will be given slowly through a tube into a vein (infusion). People will continue to receive ASP2998 until their cancer gets worse, they can't tolerate ASP2998, they start other cancer treatment, they or the doctor decides the person should stop receiving ASP2998.

ELIGIBILITY:
Inclusion Criteria:

* For the ASP2998 monotherapy dose escalation (excluding urothelial and non-small cell lung cancer (NSCLC) tumor-specific backfill participants), the following criteria apply:

  * participant has a confirmed diagnosis of locally advanced unresectable or metastatic solid tumors.
  * Participant has progressed on, is ineligible for, or has refused all available standard therapies (no limit to the number of prior treatment regimens).
  * Prior exposure to TROP2, stimulator of interferon genes (STING) agonist or topoisomerase I (TopI) directed therapy is allowed.
  * Participant must have one of the following malignancies: Urothelial carcinoma, NSCLC, Gastric/ gastroesophageal junction (GEJ) cancer, Breast cancer (human epidermal growth factor receptor 2 [HER2]-negative; local testing for HER2 status is acceptable).
  * For all tumor types, any component of neuroendocrine histology is ineligible.
* For the ASP2998 NSCLC second line (2L)+ Monotherapy Dose Expansion Cohort(s) (including the tumor-specific backfill participants from the monotherapy dose escalation), the following criteria apply:

  * Participant has locally advanced unresectable or metastatic NSCLC with known programmed cell death-1 (PD-L1) status, without actionable oncogenic alteration (AGA), according to local testing.
  * Participant must have histologically or cytologically confirmed diagnosis of locally advanced unresectable or metastatic NSCLC that has progressed on or after receiving platinum-based chemotherapy and/or checkpoint inhibitors according to local/regional standard of care.
  * Participant is also eligible if there is disease progression within 12 months of receiving neoadjuvant or adjuvant therapy for resectable disease.
  * Participant must be eligible to receive treatment in 2L+ setting.
  * Participant must have had no more than 3 prior lines of therapy.
  * No prior exposure to TROP2, STING agonist or TopI directed therapy is allowed.
* For the ASP2998 Urothelial Carcinoma Monotherapy Dose Expansion Cohort(s) (including the tumor-specific backfill participants from the monotherapy dose escalation), the following criteria apply:

  * Participant must have histologically or cytologically confirmed diagnosis of urothelial carcinoma (i.e., cancer of the bladder, renal pelvis, ureter or urethra) in locally advanced unresectable or metastatic setting that has progressed on a combination of enfortumab vedotin and pembrolizumab according to local/regional standard of care. Participant with urothelial carcinoma (transitional cell) with < 50% squamous differentiation or mixed cell types is eligible.
  * Participant is also eligible if there is disease progression within 12 months of receiving adjuvant or neoadjuvant therapy for resectable disease.
  * Participant must be eligible to receive treatment in 2L+ setting.
  * Participant must have had no more than 3 prior lines of therapy.
  * No prior exposure to TROP2, STING agonist or TopI directed therapy is allowed.
* For ASP2998 combination therapy (including the tumor-specific backfill participants from the combination therapy dose escalation), the following criteria apply for the NSCLC first line (1L) ASP2998 + Pembrolizumab + Carboplatin Dose Escalation and Expansion Cohort(s):

  * Participant has locally advanced unresectable or metastatic NSCLC (adenocarcinoma only, no mixed histology allowed), with known PD-L1 status, without AGA, according to local testing.
  * Participant is also eligible if there is disease progression > 12 months after completing adjuvant or neoadjuvant therapy for resectable disease.
  * Participant has not received prior therapy for metastatic disease.
  * No prior exposure to TROP2, STING agonist or TopI directed therapy is allowed in dose escalation or dose expansion.
* For ASP2998 combination therapy (including the tumor-specific backfill participants from the combination therapy dose escalation), the following criteria apply for the Urothelial Carcinoma 1L ASP2998 + Pembrolizumab + Enfortumab Vedotin Dose Escalation and Expansion Cohort(s):

  * Participant must have histologically or cytologically confirmed diagnosis of urothelial carcinoma (i.e., cancer of the bladder, renal pelvis, ureter or urethra) in locally advanced unresectable or metastatic setting. Participant with urothelial carcinoma (transitional cell) with < 50% squamous differentiation or mixed cell types is eligible.
  * Participant is also eligible if there is disease progression > 12 months after completing adjuvant or neoadjuvant therapy for resectable disease.
  * Participant has not received prior therapy for metastatic disease.
  * No prior exposure to TROP2, STING agonist or TopI directed therapy is allowed in dose escalation or dose expansion.
* For ASP2998 combination therapy (including the tumor-specific backfill participants from the combination therapy dose escalation), the following criteria apply for the NSCLC 2L+ ASP2998 + Pembrolizumab Dose Escalation Cohort(s):

  * Participant has locally advanced unresectable or metastatic NSCLC with known PD-L1 status, without AGA, according to local testing.
  * Participant has progressed on or after receiving platinum-based chemotherapy and/or checkpoint inhibitors according to local/regional standard of care.
  * Participant is also eligible if there is disease progression within 12 months of receiving neoadjuvant or adjuvant therapy for resectable disease.
  * Participant may be eligible to receive treatment in 2L+ setting.
  * Participant must have had no more than 3 prior lines of therapy.
  * Prior exposure to TROP2, STING agonist or TopI directed therapy is allowed.
* For ASP2998 combination therapy (including the tumor-specific backfill participants from the combination therapy dose escalation), the following criteria apply for the Urothelial Carcinoma 2L+ ASP2998 + Pembrolizumab Dose Escalation Cohort(s):

  * Participant must have histologically or cytologically confirmed diagnosis of urothelial carcinoma (i.e., cancer of the bladder, renal pelvis, ureter or urethra) in locally advanced unresectable or metastatic setting that has progressed on a combination of enfortumab vedotin and pembrolizumab according to local/regional standard of care. Participant with urothelial carcinoma (transitional cell) with < 50% squamous differentiation or mixed cell types is eligible.
  * Participant is also eligible if there is disease progression within 12 months of receiving adjuvant or neoadjuvant therapy for resectable disease.
  * Participant must be eligible to receive treatment in 2L+ setting.
  * Participant must have had no more than 3 prior lines of therapy.
  * Prior exposure to TROP2, STING agonist or TopI directed therapy is allowed.
* For ASP2998 combination therapy (including the tumor-specific backfill participants from the combination therapy dose escalation), the following criteria apply for the Urothelial Carcinoma 2L+ ASP2998 + Enfortumab Vedotin Dose Escalation Cohort(s):

  * Participant must have histologically or cytologically confirmed diagnosis of urothelial carcinoma (i.e., cancer of the bladder, renal pelvis, ureter or urethra) in locally advanced unresectable or metastatic setting that has progressed on a combination of enfortumab vedotin and pembrolizumab according to local/regional standard of care. Participant with urothelial carcinoma (transitional cell) with < 50% squamous differentiation or mixed cell types is eligible.
  * Participant is also eligible if there is disease progression within 12 months of receiving adjuvant or neoadjuvant therapy for resectable disease.
  * Participant must be eligible to receive treatment in 2L+ setting.
  * Participant must have had no more than 3 prior lines of therapy.
  * Prior exposure to TROP2, STING agonist or TopI directed therapy is allowed.
* Participant has a predicted life expectancy ≥ 12 weeks.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participant has at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participant's adverse events (AEs) (excluding alopecia) from prior anticancer therapy have improved to Grade 1 or baseline within 14 days prior to the first dose of study intervention.
* Participant has adequate organ function as indicated by laboratory values (If a participant has received a recent blood transfusion, the laboratory tests must be obtained ≥ 14 days after any blood transfusion.)
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who has a negative serum pregnancy test and confirmed not pregnant by medical interview at screening and agrees to follow the contraceptive guidance from the time of informed consent through 7 months after final study intervention administration.
* Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 7 months after final study intervention administration.
* Female participant must not donate ova starting at first administration of study intervention and throughout the investigational period and for 7 months after final study intervention administration.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 7 months after final study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 7 months after final study intervention administration.
* Male participant must not donate sperm during the treatment period and for 7 months after final study intervention administration.
* Participant agrees not to participate in another interventional study while receiving study intervention in the present study/participating in the present study (participant who is currently in the follow-up period of an interventional clinical study is allowed).

Exclusion Criteria:

* Participant weighs < 40 kg during screening.
* Participant has known active central nervous system (CNS) metastases. NOTE: A participant with CNS metastases that have been treated with surgery and/or radiation therapy, who is no longer taking pharmacologic doses of glucocorticoids and is neurologically stable, is eligible. Prophylactic use of anticonvulsants is permitted.
* Any history of recurrent Grade 3 AEs/ immune-related AEs (irAEs) or history of Grade 4 AEs/irAEs.
* Participant has active or prior autoimmune or inflammatory disorders requiring systemic anti-inflammatory or immunosuppressive therapy within the past 3 years. Participants with type 1 diabetes mellitus or endocrinopathies stably maintained on appropriate replacement therapy will not be excluded.
* Participant has uncontrolled diabetes mellitus. For cohorts receiving enfortumab vedotin, uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) of ≥ 8% or HbA1c of 7% to < 8% with associated diabetes symptoms (polyuria or polydipsia).
* Participant has leptomeningeal disease as a manifestation of the current malignancy.
* Participant has a known additional malignancy that requires active treatment, with the exception of any of the following:

  * Locally curable malignancies that have been apparently cured with no recurrence in the past 2 years.
  * Adequately treated stage I cancer from which the participant is currently in remission and has been in remission for ≥ 2 years.
  * Any other cancer from which the participant has been disease-free for ≥ 5 years.
* Participant has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of first administration of study intervention. Inhaled or topical steroids and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Participant has jaundice or known current active liver disease from any cause, including hepatitis A (hepatitis A virus (HAV) immunoglobulin M (IgM) positive, but testing for hepatitis A in screening is not required), hepatitis B (hepatis B virus (HBV) (hepatitis B surface antigen positive, or HBV DNA positive if HBsAg is negative and anti-HBs and/or anti-HBc positive)), or hepatitis C (HCV antibody positive, confirmed by HCV RNA). NOTE: screening for these infections should be conducted per local requirements.
* Participant has a known history of human immunodeficiency virus (HIV) infection with acquired immunodeficiency syndrome (AIDS)-related complications. HIV testing will be conducted per local requirements.
* Participant has clinically significant cardiac disease, defined as any of the following:

  * Clinically significant cardiac arrhythmias including bradyarrhythmia which are poorly controlled. Rate-controlled atrial fibrillation is permitted.
  * Congenital long QT syndrome.
  * corrected QT interval by Fridericia (QTcF) ≥ 470 msec at screening. Electrocardiograms (ECGs) will be performed in triplicate during screening; the average of the triplicate readings will be used in the calculation of QTc. If the QTc is prolonged in a participant with a pacemaker or a right sided bundle branch block, the participant may be enrolled. Participant with a left sided bundle branch block will be excluded.
  * History of clinically significant cardiac disease or congestive heart failure greater than New York Heart Association (NYHA) Class II or left ventricular ejection fraction (LVEF) measurement of < 50% at baseline. Participant must not have had unstable angina (symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months.
  * Uncontrolled hypertension, defined as systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg that has been confirmed by 2 successive measurements, despite optimal medical management.
  * Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before start of study intervention.
* Participant has a history of non-infectious interstitial lung disease (ILD)/pneumonitis, has current Grade ≥ 1 ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening. Participant with previously diagnosed Grade 1 radiation pneumonitis is allowed to be screened for the study. Radiation pneumonitis must be confined to the previously irradiated area of the lung and completely resolved.
* Participant has inadequate pulmonary reserve due to pulmonary, heart or other disease.
* Participant has a confirmed oxygen saturation (SpO2) < 92% at screening.
* Participant requires chronic oxygen supplementation therapy.
* Participant has evidence of structural compromise to the trachea for any reason, including underlying malignancy.
* Participant has had major surgery within 4 weeks prior to first dose of study intervention.
* Participant currently has or has a history of corneal disease or inflammation of the eye.
* Participant is at a significant risk of bleeding due to medical condition(s) or use of anticoagulants, or has a history of life-threatening bleeding (e.g., intracranial bleeding).
* Participant has current peripheral neuropathy Grade 2 or higher (specific for enfortumab vedotin or carboplatin-containing cohorts only).
* Participant has a history of Grade 2 or higher hearing loss (specific for the carboplatin-containing cohort only).
* Participant has received prior TROP2 targeting agents, STING agonists or TopI inhibitor (exception: dose escalation cohorts in monotherapy and 2L+ combination therapy).
* Participant has received prior anticancer therapy within 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study intervention.
* Participant has received prior radiation therapy within 14 days of the first dose of study intervention. Participant must have recovered from all radiation-related toxicities and not require corticosteroids. A 1-week washout is permitted for palliative radiation (≤ 3 weeks of radiotherapy) to non-CNS disease.
* Participant has an active infection requiring intravenous antibiotics within 14 days prior to study intervention.
* Participant is expected to require another form of anticancer therapy while on study intervention.
* Participant is receiving anticoagulants (vitamin K antagonists or direct oral anticoagulants) or antiplatelet agents. Low dose aspirin is allowed.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study intervention.
* Participant has any condition that makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to study intervention or any components of the formulation used.
* Participant has history of life-threatening (anaphylaxis) hypersensitivity reactions to monoclonal antibodies, bispecifics, immunomodulatory drugs or antibody-drug conjugates (ADCs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to 21 days
  A DLT is defined as any event meeting the DLT criteria occurring within 21 days of first dose on Cycle 1 Day 1 (C1D1) that cannot clearly be attributed to a cause other than ASP2998 administered in monotherapy or in combination with standard treatments.
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to 21 Months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
  A TEAE is an AE with onset at any time from first dosing until last scheduled procedure.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 21 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to 19 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 19 months
  Number of participants with potentially clinically significant ECG values.
Number of Participants with Physical Examination (PE) abnormalities and/or AEs | Up to 19 months
  Number of participants with potentially clinically significant PE values.
Number of Participants at each grade of Eastern Cooperative Oncology Group (ECOG) performance status score | Up to 19 months
  The ECOG scale will be used to assess performance status. Scores range from 0 (fully active) to 5 (dead). Negative change scores represent an improvement. Positive scores represent a decline in performance.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) of ASP2998 per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 27 months
  ORR is defined as the proportion of participants whose best overall response is rated as Complete Response (CR) or Partial Response (PR) per RECIST v1.1 as assessed by the investigator.
Duration of Response (DOR) of ASP2998 per RECIST v1.1 | Up to 27 months
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented progressive disease (PD) per RECIST v1.1 as assessed by the investigator or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) of ASP2998 per RECIST v1.1 | Up to 27 months
  DCR is defined as the proportion of participants whose best overall response is rated as CR, PR or stable disease (SD) per RECIST v1.1 as assessed by the investigator.
Progression Free Survival (PFS) per RECIST v1.1 | Up to 27 months
  PFS is defined as the time from the first dose of study intervention until the date of documented PD per RECIST v1.1 as assessed by the investigator or until death for any cause, whichever comes first.
Overall Survival (OS) | Up to 33 months
  OS is defined as the time from the first dose of study intervention until death due to any cause.
Pharmacokinetics (PK) of ASP2998 in plasma: area under the concentration-time curve at 21 days (AUC21d) | Up to 18 months
  AUC21d will be recorded from the PK plasma samples collected.
PK of ASP2998 in plasma: maximum concentration (Cmax) | Up to 18 months
  Cmax will be recorded from the PK plasma samples collected.
PK of ASP2998 in plasma: trough concentration (Ctrough) | Up to 18 months
  Ctrough will be recorded from the PK plasma samples collected.
PK of ASP2998 in plasma: time of maximum concentration (tmax) | Up to 18 months
  tmax will be recorded from the PK plasma samples collected.
Incidence rate of trophoblast cell surface antigen 2 (TROP2) expression in tumor | Up to 18 months
  Incidence rate of TROP2 expression in tumor will be evaluated from tissue samples collected.
Expression levels of TROP2 in tumor | Up to 18 months
  Expression levels of TROP2 expression in tumor will be evaluated from tissue samples collected.
Change of TROP2 expression in tumor | Up to 18 months
  Change of TROP2 expression in tumor will be evaluated from tissue samples collected.
Change in CD8 T-cell lymphocytes in paired biopsies | Up to 18 months
  Change in CD8 T-cell lymphocytes in paired biopsies will be evaluated from tissue samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- START New York Long Island, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency